CLINICAL TRIAL: NCT03684798
Title: Applying Mental Contrasting With Implementation Intentions to Prevent Relapse and Drop-out in Patients With Alcohol Use Disorders
Brief Title: Mental Contrasting With Implementation Intentions for Alcohol Use Disorders
Acronym: MCIIAUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susanne Rösner (Other)
Collaborators: University of Konstanz (Other); Zurich University of Applied Sciences (Other); New York University (Other); University of Hamburg-Eppendorf (Other)
Responsible Party: Sponsor-Investigator, Susanne Rösner, Head of Research, Forel Clinic
Organization: Forel Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1
Record Dates: First submitted 2018-08-31; First posted 2018-09-26 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Alcohol Use Disorder
Keywords: MCII; Alcohol Use Disorder; Motivation; Mental Contrasting; Implementation Intentions; Abstinence
MeSH Terms: conditions — Alcoholism | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Contrasting with Implementation Intentions (MCII) (Experimental): Mental Contrasting with Implementation Intentions (MCII) combines two methods: Mental Contrasting and Implementation Intentions.
  Mental Contrasting (MC) consists of imaging a desired future and comparing it with obstacles of the present reality (Oettingen, 2000, 2014; Oettingen, Pak, & Schnetter, 2001) in order to increase goal commitment when expectations of success are high (Gollwitzer, 2014). Implementation Intentions on the other hand specify when, where, and how to strive for a goal in form of an if-then-plan, e.g. "If situation Y is encountered, then I will perform the goal-directed response Z" (Gollwitzer, 2014; Wieber, Thürmer, & Gollwitzer, 2015).
  Interventions: Other: MCII
- Treatment as usual (Active Comparator): The control group receive a control training, which consists of an exercise from treatment as usual. Thus, patients in the control group are supported in their intention for abstinence and in the reappraisal of risk situations and relapse, while no individual motivational strategies are planned or provided
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: MCII — In this study, the research staff will work through the MCII approach with the participant as an interactive, face-to-face training. The desired future consists of imaging an abstinent life and comparing it with personally relevant obstacles. Afterwards, the most relevant obstacle will be chosen and an if-then-plan will be formed, that refers to this obstacle.
  Arms: Mental Contrasting with Implementation Intentions (MCII)
Other: Treatment as usual — The patients in the control group will receive a 2 x 2 contingency table about the disadvantages and advantages of being abstinent and of drinking. In addition, abstinence intentions of patients in the control group will also be supported and risk situations and relapse events since the last trainings will be reappraised, but without the use of MCII.
  Arms: Treatment as usual

SUMMARY:
Mental Contrasting (MC) consists of imaging a desired future and comparing it with obstacles of the present reality in order to increase goal commitment when expectations of success are high. The study aims to investigate the effects of a motivational training (Mental Contrasting with Implementation Interventions; MCII) as a therapeutic add-on to standard treatment in inpatients with Alcohol Use Disorders.

DETAILED DESCRIPTION:
Today's elaborated therapeutic interventions do not ensure sustainability of therapeutic success in alcohol-dependent patients. Thus, it is to develop and implement new therapeutic methods in order to increase regular treatment termination and continuous abstinence during treatment. Mental Contrasting (MC) consists of imaging a desired future and comparing it with obstacles of the present reality in order to increase goal commitment when expectations of success are high.

In the study, MCII is implemented as an add-on intervention in order to reduce the risk of a relapse during treatment and to decrease drop-outs from treatment in alcohol-dependent inpatients. Therefore, inpatients with alcohol use disorder (AUD) are randomly assigned to one of two groups. The experimental group does receive MCII, the control group an exercise from treatment as usual. In addition, patients undergo brief motivational screenings in form of self-report questionnaires at the beginning and during treatment in order to assess motivational mediation of treatment effects and drinking events. The effect of the MCII training will be examined on primary (drinking during treatment) and secondary outcome variables (early treatment termination, motivational changes after drinking events).

The Primary Outcome is return to drinking during treatment defined as any violation of total abstinence. Drinking is assumed if either a drinking event is reported by the patient or a Breathalyzer tests is positive.

Participants are allocated to the groups using randomisation with emphasis on equal group sizes in control and experimental group. The list of randomisation was generated with the online tool "Research Randomizer".

The investigator's a priori calculation of the required sample size is based on the primary outcome, i.e. return to any drinking during treatment. Given α=0.05 and 1-β=0.80 a one-sided z-test then yields a required sample size of 122 participants, i.e. 61 subjects in the intervention group and 61 subjects in the control group.

All randomized subjects will be included in the analyses, regardless of whether they terminate the study regularly or not. Analyses will be done according to the intention-to-treat method (ITT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcohol use disorder according to DSM 5 (Diagnostic and Statistical Manual)
* Age: ≥18 years

Exclusion Criteria:

* Cognitive deficits that limit the patients' ability to provide informed consent
* Inability to follow the procedures of the study
* Acute suicidality
* Acute psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with return to any drinking | through study completion at end of treatment, an average of 10 weeks
  Any drinking as measured by self-report or objective testing
Rate of number of drinking events during treatment | through study completion at end of treatment, an average of 10 weeks
  Drinking Events as measured by self-report

SECONDARY OUTCOMES:
Number of participants with early treatment termination | through study completion at end of treatment, an average of 10 weeks
  Treatment Termination without consent between patient and therapist
Rate of general self-efficacy for abstinence | through study completion at end of treatment, an average of 10 weeks
  self-efficacy will be assessed on the proposal of Ludwig, Tadayon-Manssuri, Strik, and Moggi (2013) to measure self-efficacy with simply one question ("How confident are you that you will be completely abstinent in 1 year, on a scale from 1 to 10?"). This scale is called "general self-efficacy". Lower scores indicate low self-efficacy and therefore a worse outcome; higher scores indicate a high self-efficacy and consequently a better outcome. We changed this question for different time intervals (e.g. the next fourteen days, until the end of treatment). The subscales are analyzed individually.
Rate of goal commitment for abstinence | through study completion at end of treatment, an average of 10 weeks
  Goal commitment will be assessed with the "Commitment to Sobriety Scale" (Kelly & Greene, 2014). It is a brief five-item measure to assess level of client commitment to alcohol and drug use cessation and continued abstinence. Each item is rated on a 6-point Likert scale from strongly disagree (1) to strongly agree (6). Lower scores indicate low commitment to sobriety and therefore a worse outcome; higher scores indicate a high commitment to sobriety and consequently a better outcome. A total score will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Rösner, Principal Investigator — Forel Clinic
Locations (1):
- Forel Klinik, Ellikon, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oettingen G. Expectancy effects on behavior depend on self-regulatory thought. Social Cognition 18(2): 101-129, 2000.
- [Background] Oettingen G. Rethinking positive thinking: inside the new science of motivation. New York, NY: Penguin Random House, 2014.
- [Background] Oettingen G, Pak H, Schnetter K. Self-regulation of goal setting: turning free fantasies about the future into binding goals. J Pers Soc Psychol. 2001 May;80(5):736-53. PMID 11374746
- [Background] Gollwitzer PM. Weakness of the will: Is a quick fix possible? Motivation and Emotion 38: 305-322, 2014.